CLINICAL TRIAL: NCT04215991
Title: An Open-label Study With a Nonrandomized Single-dose Phase in Subjects With Suspected or Confirmed Aerobic Gram-negative Bacterial Infections Followed by a Randomized, Multiple-dose, Active-controlled Phase in Subjects With Suspected or Confirmed Complicated Urinary Tract Infection (cUTI), Hospital-acquired Bacterial Pneumonia (HABP) or Ventilator-associated Bacterial Pneumonia (VABP) to Assess the Safety, Tolerability, and Pharmacokinetics of Cefiderocol in Hospitalized Pediatric Subjects 3 Months to < 18 Years of Age
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of Cefiderocol in Hospitalized Pediatric Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1704R2133; 2019-002121-30 (EudraCT Number)
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Gram-negative Bacterial Infections; Hospital Acquired Bacterial Pneumonia (HABP); Complicated Urinary Tract Infection (cUTI); Ventilator Associated Bacterial Pneumonia (VABP)
MeSH Terms: conditions — Gram-Negative Bacterial Infections | interventions — Cefiderocol; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single Dose Phase: Cefiderocol (Experimental): Participants will receive a single dose of cefiderocol administered intravenously (IV) on Day 1, in addition to standard of care. Participants weighing less than 34 kilograms (kg) will receive 60 milligrams (mg)/kg cefiderocol and participants ≥34 kg will receive 2000 mg.
  Interventions: Drug: Cefiderocol; Drug: Standard of Care
- Multiple Dose Phase: Cefiderocol (Experimental): Participants will receive cefiderocol administered via IV every 8 hours for an expected 5 to 14 days in addition to standard of care. Participants weighing less than 34 kg will receive 60 mg/kg cefiderocol and participants ≥ 34 kg will receive 2000 mg. Dosage may be adjusted based on renal function.
  Interventions: Drug: Cefiderocol; Drug: Standard of Care
- Multiple Dose Phase: Standard of Care Alone (Active Comparator): Participants will receive standard of care treatment according to local standards.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Cefiderocol — Administered intravenously over 3 hours
  Other Names: Fetroja; S-649266
  Arms: Multiple Dose Phase: Cefiderocol; Single Dose Phase: Cefiderocol
Drug: Standard of Care — Standard of care administered will be selected by the investigator based on the suspected or confirmed pathogen(s) for the infection in accordance with local standards.

SUMMARY:
The primary objectives of this study are to assess the safety, tolerability, and pharmacokinetics (PK) of cefiderocol after single-dose administration in hospitalized pediatric participants 3 months to < 12 years of age with suspected or confirmed aerobic Gram-negative bacterial infections and after multiple-dose administration in hospitalized pediatric participants 3 months to < 18 years of age with suspected or confirmed complicated urinary tract infection (cUTI), hospital-acquired bacterial pneumonia (HABP), or ventilator-associated bacterial pneumonia (VABP).

DETAILED DESCRIPTION:
This study consists of a nonrandomized single-dose phase in children aged 3 months to less than 12 years with suspected or confirmed aerobic Gram-negative bacterial infections and a randomized multiple-dose, active-comparator standard of care (SOC) phase in children aged 3 months to less than 18 years with cUTI, HABP, or VABP to assess the PK, safety, and tolerability of cefiderocol in hospitalized participants requiring systemic antibiotics for an expected 5 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Participant's parent(s) or legally authorized representative(s) (LAR) provides written informed consent in accordance with regional- and country-specific laws and regulations
2. Participant provides written informed assent, when feasible (age of assent to be determined by institutional review board/independent ethics committee [IRBs/IECs] or be consistent with local legal requirements)
3. Hospitalized participant is 3 months to < 18 years of age at the time written informed consent/assent is obtained for the multiple-dose phase. Hospitalized participant is 3 months to < 12 years of age at the time written informed consent/assent is obtained for the single-dose phase.
4. Single-dose phase: Participant has a suspected or confirmed infection type (including but not limited to cUTI, complicated intra-abdominal infections [cIAI], pneumonia, HABP/VABP, and sepsis or bloodstream infections [BSI]) that requires hospitalization for treatment with IV antibiotics.

   Multiple-dose phase: Participant has a suspected or confirmed cUTI, HABP, or VABP that requires hospitalization for treatment with IV antibiotics
5. If participant is a sexually active female of childbearing potential and has reached menarche or Tanner stage 3, participant agrees to use barrier contraception (including condom, diaphragm, or cervical cap) with spermicide or agrees to use a highly effective method of contraception (including contraceptive implant, injectable contraceptive, combination oral contraceptive, or an intrauterine [IUD] contraceptive device) from Screening up to 28 days after administration of the last dose of cefiderocol.

Exclusion Criteria:

1. Participant has a documented history of any hypersensitivity or allergic reaction to any β-lactam antibiotic (Note: for β-lactams, a history of a mild rash followed by uneventful re-exposure is not a contraindication to enrollment.)
2. Multiple-dose only: Participant has an infection caused only by a confirmed Gram-positive pathogen.
3. Participant has a suspected or confirmed central nervous system (CNS) infection (for example, meningitis, brain abscess, shunt infection) or osteomyelitis (which would require prolonged antibiotic therapy).
4. Participant has cystic fibrosis.
5. Single-dose phase: Participant has moderate or severe renal impairment based on estimated glomerular filtration rate (eGFR) (based on the Schwartz equation if ≥ 3 months to < 1 year of age and modified Bedside Schwartz equation if ≥ 1 to < 18 years of age) of < 60 milliliter (mL)/ minute (min)/1.73 square meters (m^2)² at Screening .

   Multiple-dose phase: Participant has an eGFR (based on the Schwartz equation if ≥ 3 months to < 1 year of age and modified Bedside Schwartz equation if ≥ 1 to < 18 years of age) of < 15 mL/min/1.73 m² at Screening.
6. Participant has end-stage renal disease (ESRD), is on hemodialysis (HD), or receiving continuous venovenous hemofiltration (CVVH).
7. Participant has experienced shock in the prior month or is in shock at the time of Screening.
8. Participant has severe neutropenia or is severely immunocompromised.
9. Participant has multiorgan failure .
10. Participant with a life expectancy of < 30 days due to severity of a concurrent illness.
11. Participant is a female who has a positive pregnancy test at Screening.
12. Participant is a female who is breastfeeding.
13. Participant has received any other investigational medicinal product (IMP) within 30 days.
14. Participant has any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data, including acute trauma to the pelvis or urinary tract.
15. Participant is receiving vasopressor therapy at Screening.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events in the Single Dose Phase | 28 days
Maximum Observed Plasma Concentration (Cmax) of Cefiderocol in the Single Dose Phase | Day 1, 1 (cohort 2 only), 3, 3.5 (cohort 2 only), 5, and 8 hours after the start of infusion
Area Under the Plasma Concentration Time Curve Extrapolated from Time 0 to Infinity (AUCinf) of Cefiderocol in the Single Dose Phase | Day 1, 1 (cohort 2 only), 3, 3.5 (cohort 2 only), 5, and 8 hours after the start of infusion
Apparent Terminal Elimination Half-life of Cefiderocol in the Single Dose Phase | Day 1, 1 (cohort 2 only), 3, 3.5 (cohort 2 only), 5, and 8 hours after the start of infusion
Number of Participants with Adverse Events in the Multiple Dose Phase | Up to 28 days after last dose (33 to 42 days depending on treatment duration)
Maximum Observed Plasma Concentration of Cefiderocol in the Multiple Dose Phase | During one of the dosing intervals from Day 5-14, 1 (cohort 2 1 and 2 only), 3, 3.5 (cohorts 1 and 2 only), 5, and 8 hours after the start of infusion
Area Under the Plasma Concentration Time Curve Over the Dosing Interval τ (AUC0-τ) of Cefiderocol in the Multiple Dose Phase | During one of the dosing intervals from Day 5-14, 1 (cohort 2 1 and 2 only), 3, 3.5 (cohorts 1 and 2 only), 5, and 8 hours after the start of infusion
Apparent Terminal Elimination Half-life of Cefiderocol in the Multiple Dose Phase | During one of the dosing intervals from Day 5-14, 1 (cohort 2 1 and 2 only), 3, 3.5 (cohorts 1 and 2 only), 5, and 8 hours after the start of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (25):
- United States (2):
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Cook Children's Medical Center, Fort Worth, Texas
- Queensland Children's Health Precinct Level 8, Centre for Children's Health Research 62 Graham Street, South Brisbane, Queensland, Australia
- Georgia (2):
  - JSC "EVEX Medical Corporation"- M Lashvili Childrens Central Hospital, Tbilisi
  - Ltd Unimedi Kakheti Childrens New Clinic, Tbilisi
- Greece (5):
  - Heraklion University General Hospital, Heraklion, Crete
  - University General Hospital of Larissa, Larissa, Thessaly
  - University Hospital "ATTIKON" 3rd Pediatric Clinic of NKUA, Chaïdári
  - Hippokration Hospital 3rd Pediatric Clinic of AUTH Konstantinoupoleos 49, Thessaloniki
  - General Hospital of Thessaloniki Papageorgiou, Thessaloniki
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Klaipeda Children's Hospital, Klaipėda
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Mexico (2):
  - Hospital Civil de Guadalajara Hospital 278, El retiro, Torre Piso 10, Infectología Ped., Guadalajara, Jalisco
  - Instituto Nacional de Pediatría "Laboratorio de la Unidad de Apoyo a la Investigación Clínica", Planta Baja Col. Insurgentes Cuicuilco, Delegacion Coyoacán Av. Insurgentes Sur 3700-C, Mexico City
- Panama (2):
  - Hospital de Especialidades Ped Via España y Calle Zarak, Panama City
  - Hospital del Niño, Epidemiologia, Panama City
- Philippines (3):
  - Chong Hua Hospital, Cebu City
  - Western Visayas and Medical Center, Iloilo City
  - Manila Doctor's Hospital, Manila
- Spain (2):
  - Hospital Val d'Hebron, Barcelona
  - Hospital del Mar, Passeig Marítim 25-29, Barcelona
- Ukraine (3):
  - Municipal Noncommercial Enterprise of Kharkiv Regional Council " V.I.Shapoval Regional Clinical Center of Urology and Nephrology", Department of Children Urology # 7, Kharkiv
  - Vinnytsia Regional Children's Hospital, Vinnytsia
  - Zaporizhzhia Regional Children Clinical Hospital, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bradley JS, Orchiston E, Portsmouth S, Ariyasu M, Baba T, Katsube T, Makinde O. Pharmacokinetics, Safety and Tolerability of Single-dose or Multiple-dose Cefiderocol in Hospitalized Pediatric Patients Three Months to Less Than Eighteen Years Old With Infections Treated With Standard-of-care Antibiotics in the PEDI-CEFI Phase 2 Study. Pediatr Infect Dis J. 2025 Feb 1;44(2):136-142. doi: 10.1097/INF.0000000000004529. Epub 2024 Sep 4. PMID 39230271